CLINICAL TRIAL: NCT03825874
Title: Comparison of the Impact on Digestive Portage of Broad Spectrum Beta-Lactamase-Producing Enterobacteriaceae (E-ESBLs) of Proposed Treatments in Outbreaks of Childhood Urinary Tract Infection
Brief Title: Research of the Consequences on the Digestive Tract Following the Proposed Treatments for a Urinary Infection in Children
Acronym: MIKA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: MIKA; 2017-A02372-51 (Other: ID-RCB)
Record Dates: First submitted 2018-08-08; First posted 2019-01-31 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Urinary Tract Infections; Urinary Tract Infections in Children
MeSH Terms: conditions — Urinary Tract Infections | interventions — Amikacin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — anorectal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- amikacin IV: Febrile urinary tract infection treated with amikacin IV
  Interventions: Other: Amikacin
- Other antibiotics: Febrile urinary tract infection treated with other antibiotic, according to the recommendations: ceftriaxone or cefixime
  Interventions: Other: usual antibiotic treatment

INTERVENTIONS:
Other: Amikacin — A first anorectal swab will be performed before starting any antibiotic treatment Three to four days after the start of antibiotic treatment, patients will be seen again and a new anorectal swab will be performed.
  Groups: amikacin IV
Other: usual antibiotic treatment — A first anorectal swab will be performed before starting any antibiotic treatment Three to four days after the start of antibiotic treatment, patients will be seen again and a new anorectal swab will be performed.
  Groups: Other antibiotics

SUMMARY:
The emergence of extended-spectrum beta-lactamase-producing Enterobacteriaceae (E-ESBL) is a major public health problem. It leads more frequent prescription of penems with the risk of emergence and spread of strains producing carbapenemases, which may be resistant to all known antibiotics. A policy of savings of penems is desirable. Among the alternatives to penems, amikacin is in the foreground. It remains active on the majority of E-ESBL strains. Some risk factors for E-ESBL emergence are known: recent antibiotic therapy (particularly quinolones and cephalosporins third generation), previous hospitalization or residence in a high endemic country.

In pediatrics, E-ESBLs are primarily responsible for urinary tract infection. In France, E-ESBLs represent about 10% of the strains responsible for urinary tract infections. The Pathology Group Pediatric Infectious (GPIP) of the French Society of Pediatrics (SFP) and the Society of Infectious Pathology French Language (SPILF) have proposed different therapeutic options to treat febrile UTIs in children: amikacin intravenous; intravenous (IV) ceftriaxone or intramuscular (IM); or cefixime per-os (PO).

The objective of this study is to compare the emergence of E-ESBLs in stools of children after febrile UTIs treatment with amikacin IV versus ceftriaxone or cefixime.

ELIGIBILITY:
Inclusion Criteria:

* Infant and child (age ≥ 3 months and <3 years)
* Patient treated for febrile urinary tract infection as monotherapy with amikacin IV, ceftriaxone (IV or IM) or cefixime PO *
* Whose parents read and understood the newsletter and whose express consent was collected
* Patient affiliated to a social security scheme (Social Security or Universal Medical Coverage)

Exclusion Criteria:

* Child treated with more than one antibiotic (eg treatment with dual therapy ceftriaxone / cefotaxime and aminoglycoside)
* Antibiotherapy in progress or discontinued in the previous 7 days
* Hospitalized child
* Refusal of one of the parents

Ages: 3 Months to 3 Years | Sex: All
Age Groups: Child
Study Population: Child from 3 months to 3 years treated for febrile urinary tract infection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Presence of E-BLSE in stools | day 4
  ano-rectal swab

SECONDARY OUTCOMES:
Type of E-BLSE strain in stools | day 4
Rate of enzymatic resistance of E-BLSE strain in stools | 4 days
Fever | 4 days
  Time of apyrexia
side effects due to antibiotic therapy | at 1.5 months
rate of relapse of urinary tract infection | 1.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Fouad MADHI, MD, Principal Investigator — CHI Créteil
Locations (20):
- France (20):
  - Cabinet du Dr Benali, Charenton-le-Pont
  - Cabinet du Dr Coicadan, Chennevières-sur-Marne
  - Cabinet du Dr Corrard, Combs-la-Ville
  - Cabinet du Dr Thollot, Essey-lès-Nancy
  - CHU Le Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - 157 Avenue du Général Leclerc, Maisons-Alfort
  - Centre Hospitalier de Meaux, Meaux
  - Cabinet du Dr Deberdt, Nogent-sur-Marne
  - Cabinet du Dr Wollner, Nogent-sur-Marne
  - Cabinet du Dr Romain, Paris
  - Cabinet du Dr Turberg-Romain, Paris
  - Cabinet du Dr Michot, Paris
  - Hospital Robert-Debré, Paris
  - Cabinet du Dr Cohen, Saint-Maur-des-Fossés
  - Cabinet du Dr Werner, Villeneuve-lès-Avignon
  - CHI Villeneuve-Saint-Georges, Villeneuve-Saint-Georges
  - 13 Villa Beauséjour, Vincennes
  - Jean Verdier Hospital, Bondy, Île-de-France Region
  - Antoine Beclère Hospital, Clamart, Île-de-France Region
  - André Mignot Hospital, Le Chesnay, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No